CLINICAL TRIAL: NCT03247829
Title: Investigation to Optimize Hemodynamic Management of HeartMate II™ Left Ventricular Assist Device Patients Using the CardioMEMS™ Pulmonary Artery Pressure Sensor in Advanced Heart Failure
Brief Title: Investigation to Optimize Hemodynamic Management of Left Ventricular Assist Devices Using the CardioMEMS™
Acronym: INTELLECT 2-HF
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10178
Record Dates: First submitted 2017-08-04; First posted 2017-08-14 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: CardioMEMS; Left Ventricular Assist Device; Hemodynamic Management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients with CardioMEMS PA Sensor and HeartMate LVAD prior to study enrollment: Patients with CardioMEMS PA Sensor and LVAD, previously implanted, will receive hemodynamic management using CardioMEMS HF System
  Interventions: Device: Hemodynamic management using CardioMEMS HF System
- Group B: Patients with existing HeartMate LVAD implanted with CardioMEMS PA Sensor post enrollment: Patients with a HeartMate LVAD prior to study enrollment who are implanted with a CardioMEMS PA Sensor within 72 hours of study enrollment, will receive hemodynamic management using CardioMEMS HF System
  Interventions: Device: Hemodynamic management using CardioMEMS HF System

INTERVENTIONS:
Device: Hemodynamic management using CardioMEMS HF System — Using the CardioMEMS HF System, clinicians will treat to target PA pressure ranges

SUMMARY:
This observational post market study is intended to characterize hemodynamic-guided management of patients with an existing left ventricular assist device (LVAD) to protocol specified target ranges and its impact on functional status, quality of life, and readmissions

DETAILED DESCRIPTION:
The study is an observational, single group study where all participants receive the same intervention. The study plans to enroll up to 100 patients at 25 US sites. All patients will have a HeartMate Left Ventricular Assist Device (LVAD) and a CardioMEMS device implanted as standard of care. After enrollment into the study, the patient will be followed until six month follow up completion. The objective of this clinical investigation is to understand the role of hemodynamic monitoring in LVAD patients and:

* Characterize PA pressure measurements with the CardioMEMS HF System in LVAD patients under different clinical and physiologic conditions
* Characterize the effects of PA pressure on functional status, quality of life, and hospital readmissions of LVAD patients
* Evaluate target ranges for PA pressure and assess the impact of medication and pump speed changes on PA pressures

ELIGIBILITY:
Inclusion Criteria:

1. Subject has CardioMEMS HF PA Sensor and a commercially-approved HeartMate LVAD (Group A) OR Subject has commercially-approved HeartMate LVAD, is experiencing NYHA class III symptoms, and has had a previous HF hospitalization and meets FDA indications for CardioMEMS. The CardioMEMS PA Sensor must be implanted within 72 hours of consent (Group B)
2. Signed an informed consent form and agreed to provide access to patient and device data (including CardioMEMS Merlin.net data)
3. No connectivity or transmission problems with CardioMEMS
4. On HeartMate LVAD support for at least 3 months
5. Age ≥ 18 years

Exclusion Criteria:

1. Current participation in an investigation that is likely to confound study results or affect study outcome
2. Current participation in the MOMENTUM3 IDE Clinical trial and has not completed the two year follow-up for that trial
3. Inability to perform 6MHW test due to conditions other than heart failure (e.g. severe arthritis, orthopedic issues, amputation etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure patients will be recruited from the clinicians practice based on the presence of both devices under study
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sundareswaran, Study Director — Abbott
Locations (23):
- United States (23):
  - Scripps Health, La Jolla, California
  - USC University Hospital, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - San Diego Cardiac, San Diego, California
  - California Pacific Medical Center - Van Ness Campus, San Francisco, California
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - The Nebraska Medical Center, Omaha, Nebraska
  - North Shore University Hospital, Manhasset, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of North Carolina, Raleigh, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sate University, Columbus, Ohio
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Palmetto Health Richland, Columbia, South Carolina
  - The Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Aurora Medical Center, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thohan V, Abraham J, Burdorf A, Sulemanjee N, Jaski B, Guglin M, Pagani FD, Vidula H, Majure DT, Napier R, Heywood TJ, Cogswell R, Dirckx N, Farrar DJ, Drakos SG; INTELLECT 2-HF Investigators. Use of a Pulmonary Artery Pressure Sensor to Manage Patients With Left Ventricular Assist Devices. Circ Heart Fail. 2023 Jun;16(6):e009960. doi: 10.1161/CIRCHEARTFAILURE.122.009960. Epub 2023 Apr 20. PMID 37079511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 101 subjects at 22 investigational sites in the United States. The first subject was enrolled on 24 August 2017 and enrollment was completed on 20 August 2019. The last 6-month follow-up was completed on 6 March 2020. Data was collected until the database closure date, 3 April 2020.
Groups:
- Group A: Patients with both a CardioMEMS PA Sensor and HeartMate II or HeartMate 3 Left Ventricular Assist Device (LVAD) previously implanted, will receive hemodynamic management guided using hemodynamic data as measured by the CardioMEMS HF System
- Group B: Patients with a HeartMate II or HeartMate 3 LVAD previously implanted who are implanted with a CardioMEMS PA Sensor within 72 hours of enrollment, will receive hemodynamic management guided using hemodynamic data as measured by the CardioMEMS HF System.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 53 | 48
Completed | 46 | 42
Not Completed | 7 | 6
Not completed — Death | 3 | 4
Not completed — Enter Hospice Care | 1 | 0
Not completed — LVAD System Replaced / Exchange | 1 | 0
Not completed — LVAD Explant | 1 | 1
Not completed — Transplant | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group A: Patients with CardioMEMS and LVAD, previously implanted, will receive hemodynamic management using CardioMEMS
  Hemodynamic management using CardioMEMS: Using the CardioMEMS HF system, clinicians will treat to target PA pressure ranges
- Group B: Patients with LVAD to implant CardioMEMS device within 72 hours of enrollment, will receive hemodynamic management using CardioMEMS
  Hemodynamic management using CardioMEMS: Using the CardioMEMS HF system, clinicians will treat to target PA pressure ranges.
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 53 | 48 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (11.4) | 59.9 (13.6) | 61.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 39 | 37 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 53 | 48 | 101
Ischemic Cardiomyopathy [Count of Participants; unit: Participants] | 25 | 22 | 47
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.31 (7.78) | 34.08 (7.52) | 33.15 (7.67)
Systemic Systolic Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Systemic Systolic Pressure was not acquired from all patients at baseline.
  mmHg
    number analyzed (Participants) | 19 | 23 | 42
    (all) | 100.6 (30.4) | 105.7 (14.9) | 103.4 (23.1)
Systemic Diastolic Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Systemic Diastolic Pressure was not acquired from all patients at baseline.
  mmHg
    number analyzed (Participants) | 18 | 23 | 41
    (all) | 64.7 (26.6) | 72.6 (20.3) | 69.1 (23.3)
Heart Rate [Mean (Standard Deviation); unit: beats per minute] — Population: Heart Rate was not acquired from all patients at baseline.
  beats per minute
    number analyzed (Participants) | 52 | 48 | 100
    (all) | 79.2 (17.8) | 78.6 (16.1) | 78.9 (16.9)
NYHA Functional Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Functional Classification stratifies patients' heart failure (HF) by the severity of their symptoms.
  I - No limitation of physical activity. II - Slight limitation of physical activity. Comfortable at rest. III - Marked limitation of physical activity. Comfortable at rest. IV - Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  Participants
    NYHA Class I | 2 | 0 | 2
    NYHA Class II | 19 | 6 | 25
    NYHA Class III | 28 | 42 | 70
    NYHA Class IV | 4 | 0 | 4
Six Minute Walk Distance [Mean (Standard Deviation); unit: meters] — Population: Six Minute Hall Walk was not acquired from all patients at baseline.
  meters
    number analyzed (Participants) | 53 | 45 | 98
    (all) | 252.08 (136.17) | 243.76 (109.58) | 248.26 (124.11)
EQ-5D-5L VAS [Mean (Standard Deviation); unit: score on a scale] — The EQ-5D-5L self-reported questionnaire includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher quality of life. Population: EQ-5D-5L VAS test was not obtained from all patients at baseline.
  score on a scale
    number analyzed (Participants) | 53 | 46 | 99
    (all) | 70.3 (19.1) | 66.2 (20.6) | 68.4 (19.8)

OUTCOME MEASURES:

1. Primary Outcome: Six Minute Hall Walk (6MHW) Distance
Description: Change in 6MHW distance compared to baseline. The six-minute hall walk (6MHW) test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Time Frame: Six Months
Population: Six minute hall walk distance measured at 6 months compared to baseline.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Group A: Group A: Patients with CardioMEMS PA Sensor and HeartMate LVAD prior to study enrollment.
  Patients with CardioMEMS PA Sensor and LVAD, previously implanted, received hemodynamic management using CardioMEMS HF System.
- Group B: Group B: Patients with existing HeartMate LVAD at enrollment who were implanted with CardioMEMS PA Sensor post enrollment.
  Patients with a HeartMate LVAD prior to study enrollment who are implanted with a CardioMEMS PA Sensor within 72 hours of study enrollment, received hemodynamic management using CardioMEMS HF System.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 46 | 42
meters | -44.9 (135.0) | 69.7 (100.6)
Statistical Analysis 1: Comparison: Group B; Test type: Other; p = 0.001, t-test, 2 sided; Comparative p-values were calculated by two-sided t-tests (paired analysis)

2. Other Pre Specified Outcome: Change in PA Diastolic Pressure From Baseline to 6 Months
Description: Changes in PA diastolic pressure measurement over time from baseline to 6 months follow-up.
Time Frame: six months
Population: Change in PA Diastolic pressure from baseline to 6 months.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Group A | Group B
Number analyzed (Participants) | 37 | 33
mmHg | 0.6 (4.2) | -1.7 (5.6)
Statistical Analysis 1: Comparison: Group B; Test type: Other; p = 0.0931, t-test, 2 sided

3. Other Pre Specified Outcome: Days PA Diastolic Pressure is in the Pre-specified Target Range
Description: Average number of days PA diastolic pressure was in the pre-specified target range of 8-15 mmHg. For this measure, both arms were combined to assess the mean number of days, all study subjects spent in the target PA diastolic range. This was pre-defined as a whole population analysis.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: days
Groups:
- All Patients: All patients enrolled in the study.
  Hemodynamic management using CardioMEMS: Using the CardioMEMS HF system, clinicians will treat to target PA pressure ranges
Arm/Group | All Patients
Number analyzed (Participants) | 101
days | 28.2 (39.0)

4. Other Pre Specified Outcome: PA Diastolic Pressure Before 6MHW Test to After 6MHW Test
Description: Pulmonary Artery Diastolic Pressure collected using the CardioMEMS-HF system before and after the 6MHW test.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Group A Pre 6MHW Test; Group A Post 6MHW Test: Group A: Patients with CardioMEMS PA Sensor and HeartMate LVAD prior to study enrollment.
  Patients with CardioMEMS PA Sensor and LVAD, previously implanted, received hemodynamic management using CardioMEMS HF System.
- Group B Pre 6MHW Test; Group B Post 6MHW Test: Group B: Patients with existing HeartMate LVAD at enrollment who were implanted with CardioMEMS PA Sensor post enrollment.
  Patients with a HeartMate LVAD prior to study enrollment who are implanted with a CardioMEMS PA Sensor within 72 hours of study enrollment, received hemodynamic management using CardioMEMS HF System.
Arm/Group | Group A Pre 6MHW Test | Group A Post 6MHW Test | Group B Pre 6MHW Test | Group B Post 6MHW Test
Number analyzed (Participants) | 44 | 39 | 38 | 35
mmHg | 13.9 (7.2) | 16.3 (6.8) | 15.8 (8.2) | 19.8 (10.6)

5. Other Pre Specified Outcome: Number of Subjects With Either CardioMEMS or HeartMate Device Malfunctions
Description: Loss of performance, such as inability to submit pressure data for CardioMEMS and/or Pump failure for LVAD. This measure is independent of study arm as both patients had both devices at enrollment. This was pre-defined as a whole population analysis.
Time Frame: six months
Population: All patients with LVAD and CardioMEMS device in place.
Measure: Count of Participants; unit: Participants
Groups:
- All Patients: All patients with an LVAD and CardioMEMS device in place.
Arm/Group | All Patients
Number analyzed (Participants) | 101
Participants
  No Device Malfunction (HM II & HM3) | 99
  Pump thrombosis (HM II) | 1
  Driveline fracture (HM II) | 1

6. Other Pre Specified Outcome: New York Heart Association (NYHA) Classification
Description: Change in NYHA classification from baseline assessed at 6 months. New York Heart Association (NYHA) Functional Classification stratifies patients' heart failure (HF) by the severity of their symptoms.
  I - No limitation of physical activity. II - Slight limitation of physical activity. Comfortable at rest. III - Marked limitation of physical activity. Comfortable at rest. IV - Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
Time Frame: six months
Population: NYHA class as a continuous variable in which the change in NYHA class is calculated using: NYHA class I =1, class II = 2, class IIIa/IIIb = 3, class IV = 4 and death =5.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in NYHA Class
Arm/Group | Group A | Group B
Number analyzed (Participants) | 53 | 48
Change in NYHA Class | 0.12 [-0.11 to 0.35] | -0.10 [-0.32 to 0.11]

7. Other Pre Specified Outcome: EQ-5D-5L VAS
Description: Health related quality of life (EQ-5D-5L). The EQ-5D-5L self-reported questionnaire includes a visual analog scale (VAS), which records the respondent's self-rated health status on a graduated (0-100) scale, with higher scores for higher quality of life. For this measure, both arms were combined to assess the mean of and changes to the EQ-5D-5L VAS for all study subjects, as all subjects were treated the same and had the same devices once enrolled. This was pre-defined as a whole population analysis.
Time Frame: six months
Population: Change in EQ-5D-5L VAS scores from baseline to 6 months.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in score
Arm/Group | Group A | Group B
Number analyzed (Participants) | 53 | 48
Change in score | -1.4 [-7.7 to 4.9] | 3.0 [-3.2 to 9.1]

8. Other Pre Specified Outcome: Number and Percent of Participants With All-cause Hospitalizations.
Description: Number and percent of participants who were hospitalized for any cause during follow-up.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 53 | 48
Participants | 27 | 25

9. Other Pre Specified Outcome: Number and Percent of Participants With Worsening Heart Failure Events
Description: Worsening HF events incudes emergency department visits, or unscheduled clinic visits for worsening HF, volume management, and/or cardiovascular medication management.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 53 | 48
Participants | 10 | 14

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- All Patients: Patients with both an LVAD and CardioMEMS device in place. All safety assessments were made on a population basis, as all subjects were treated the same and had the same devices once enrolled. This was pre-defined as a whole population analysis.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 7/101
Serious Adverse Events (participants affected / at risk) | 36/101
Other Adverse Events (participants affected / at risk) | 3/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=101)
Worsening Heart Failure (Cardiac disorders) | 20 (23) — Worsening Heart Failure
Syncope/presyncope/dizziness and hypovolemia (Cardiac disorders) | 11 (14) — Syncope/presyncope/dizziness and hypovolemia
Cardiac arrhythmias (Cardiac disorders) | 5 (6) — Cardiac arrhythmias
Right heart failure (Cardiac disorders) | 5 (5) — Right heart failure
Renal dysfunction secondary to heart failure (Renal and urinary disorders) | 3 (4) — Renal dysfunction secondary to heart failure
Other neurological event (Nervous system disorders) | 2 (2) — Other neurological event
Respiratory failure secondary to cardiovascular cause (Vascular disorders) | 1 (1) — Respiratory failure secondary to cardiovascular cause
Strokes regardless of their type and etiology (Nervous system disorders) | 1 (1) — Strokes regardless of their type and etiology
Other (General disorders) | 4 (5) — Other
Pneumonia (Infections and infestations) | 1 (2) — Pneumonia
Hypotension (Cardiac disorders) | 1 (1) — Hypotension
Over-diuresis (Renal and urinary disorders) | 1 (1) — Over-diuresis
Volume Overload (Cardiac disorders) | 1 (1) — Volume Overload
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=101)
Non-serious Adverse Device Effects (Cardiac disorders) | 3 (3) — Events were classified by organ class only for non-serious adverse device effects.

LIMITATIONS AND CAVEATS:
No limitations or caveats to disclose for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03247829/Prot_SAP_ICF_000.pdf